CLINICAL TRIAL: NCT03287414
Title: A Subject-, Investigator-, and Sponsor-blinded, Randomized, Placebo-controlled, Multicenter Study to Investigate Efficacy, Safety, and Tolerability of VAY736 in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Study of Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of VAY736 in Patients With Idiopathic Pulmonary Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736X2207; 2017 002667 17 (EudraCT Number)
Record Dates: First submitted 2017-09-12; First posted 2017-09-19 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis; VAY736
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — ianalumab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VAY736 (Experimental): Participants received 300 mg VAY736 administered subcutaneously every 4 weeks for 48 weeks on top of current standard-of-care therapy
  Interventions: Drug: VAY736; Drug: Standard of Care (SoC)
- Placebo (Placebo Comparator): Participants received placebo administered subcutaneously every 4 weeks for 48 weeks on top of current standard-of-care therapy
  Interventions: Drug: Placebo; Drug: Standard of Care (SoC)

INTERVENTIONS:
Drug: VAY736 — 300 mg VAY736 administered subcutaneously every 4 weeks for 48 weeks
  Other Names: Ianalumab
  Arms: VAY736
Drug: Placebo — Placebo administered subcutaneously every 4 weeks for 48 weeks
  Arms: Placebo
Drug: Standard of Care (SoC) — Background standard-of-care treatment for IPF: nintedanib, pirfenidone, or no background therapy

SUMMARY:
The purpose of this study was to investigate the safety, tolerability and efficacy of VAY736 as potential therapy for the treatment of idiopathic pulmonary fibrosis (IPF).

DETAILED DESCRIPTION:
This was an exploratory (non-confirmatory) randomized, patient-, investigator-, sponsor- blinded, placebo controlled study of VAY736 in IPF patients. This study investigated the safety and efficacy of 300 mg VAY736 administered subcutaneously (s.c.) every 4 weeks for 48 weeks.

Participants were randomized in a 1:1 ratio on top of local standard of care (SOC), to receive VAY736 or placebo. Randomized subjects entered the treatment epoch (for up to 48 weeks), followed by two follow-up epochs: the PK/safety follow-up epoch and the PD/safety follow-up epoch. The PK/safety follow-up epoch lasted for 20 weeks. When the PK/safety follow-up epoch was completed, participants in the placebo arm were discharged from the study; but participants in the active arm (those who had received VAY736) continued into the PD/safety follow-up epoch. Participants in the PD/safety follow-up epoch were followed until B-cell recovery (in the peripheral blood), defined as: B cells >=50/μL or B cells >= 80% of baseline (whichever occurred first). If a participant had not recovered his/her B-cells after a period of 2 years from the last dose of VAY736, then this participant was discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of definite or probable IPF within 5 years of the screening visit
* Forced Vital Capacity (FVC) 40-90% predicted (inclusive)
* Diffusing Capacity of the Lungs (DLCO), corrected for hemoglobin, 25-79% predicted (inclusive)
* Forced Expiratory Volume in first second (FEV1)/FVC >70%
* Unlikely to die from cause other than IPF within the next 3 years, in the opinion of the investigator
* Unlikely to undergo lung transplantation during this trial

Exclusion Criteria:

* Emphysema > fibrosis on screening high-resolution computed tomography (must be confirmed by central reader)
* History of major organ, hematopoietic stem cell or bone marrow transplant
* Clinically diagnosed acute exacerbation of idiopathic pulmonary fibrosis (AE-IPF) or other significant clinical worsening within 3 months of randomization
* New York Heart Association (NYHA) class III/IV Congestive Heart Failure (CHF), Ejection Fraction (EF) <25%
* Current smoker
* Prior use of any B-cell depleting therapy (e.g., rituximab, ofatumumab, or other anti-CD20 mAb, anti-CD40, anti-CD19,anti-CD22 mAb, anti-CD52 mAb, or anti-BAFF mAb)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (7):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Salt Lake City, Utah
- Novartis Investigative Site, Calgary, Alberta, Canada
- Germany (2):
  - Novartis Investigative Site, Coswig
  - Novartis Investigative Site, Hanover
- Novartis Investigative Site, Dublin, Ireland
- Italy (3):
  - Novartis Investigative Site, Forlì, FC
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Siena, SI
- United Kingdom (2):
  - Novartis Investigative Site, Cambridge, Cambridgeshire
  - Novartis Investigative Site, High Heaton, Newcastle Upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 16 centers in 6 countries.
Pre-assignment Details: A total of 142 participants were screened of which 30 participants were randomized. 1 participant in the VAY736 arm did not receive treatment as the patient withdrew consent before first dosing. Treatment epoch (duration of up to 48 weeks) was followed by: i) PK/safety follow-up epoch with duration of 20 weeks, and ii) PD/safety follow-up (only for participants who had received VAY736) until participants met pre-specified criteria for B-Cell recover or up to 2 years from the last dose of VAY736.
Period: Treatment Epoch
Arm/Group | VAY736 | Placebo
Started | 14 | 16
Treated | 13 | 16
Completed | 6 | 12
Not Completed | 8 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Study terminated by sponsor | 2 | 2
Not completed — Subject/Guardian decision | 4 | 0
Not completed — Discontinued early with reason "other" selected | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: PK/Safety Follow-up Epoch
Arm/Group | VAY736 | Placebo
Started | 7 | 13
Completed | 7 | 13
Not Completed | 0 | 0
Period: PD/Safety Follow-up Epoch
Arm/Group | VAY736 | Placebo
Started | 7 | 0
Completed | 5 | 0
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject/Guardian decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for all participants who received at least one dose of any study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | VAY736 | Placebo | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.7 (9.30) | 68.3 (8.15) | 68.9 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 12 | 15 | 27
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment Epoch (48 Weeks of Treatment) in Forced Vital Capacity (FVC).
Description: FVC was defined as the maximum amount of air that an individual was able to forcibly exhale from his / her lungs after taking the deepest breath they could. Change from baseline to end of treatment epoch (48 weeks of treatment) in Forced Vital Capacity (FVC) was analyzed using a Mixed Effects Model for Repeated Measures (MMRM) and considering all assessments collected during the treatment epoch. The model included treatment and visit as fixed effects, standard of care treatment (Nintedanib, Pirfenidone, or no treatment) as factor and baseline value as a covariate, treatment-by-visit and baseline-by-visit as interaction terms. A positive change from baseline indicates improvement. Baseline was defined as the last available assessment pre-dose before or on randomization date.
Time Frame: From baseline up to 48 weeks post first dose of study treatment
Population: Pharmacodynamic (PD) analysis set including participants with available PD data and no protocol deviations with relevant impact on PD data. Only participants with a value at both Baseline and end of treatment (48 weeks post-first dose of treatment) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liter (L)
Arm/Group | VAY736 | Placebo
Number analyzed (Participants) | 3 | 7
Liter (L) | 0.039 (0.1116) | -0.023 (0.0773)
Statistical Analysis 1: Comparison: VAY736 vs Placebo; Test type: Superiority; p = 0.3248, MMRM — 1-sided p-values were obtained using MMRM Model; Least Squares Mean Difference = 0.063, 80% CI 2-sided [-0.115 to 0.241], Standard Error of Mean 0.1379

2. Secondary Outcome: Percentage of Participants With All-cause Mortality Events
Description: All-cause mortality events were defined as deaths due to any cause. Kaplan-Meier estimates of the percentage of participants with the event of interest along with 80% two-sided confidence intervals using Greenwood's formula are provided.
Time Frame: Up to 48 weeks post first dose of study treatment
Population: PD analysis set including participants with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | VAY736 | Placebo
Number analyzed (Participants) | 12 | 16
Percentage of participants | 8.3 [2.39 to 26.92] | 0 [NA to NA] — NA: Not estimable because no events occurred within this group
Statistical Analysis 1: Comparison: VAY736 vs Placebo; Test type: Other; p = 0.868, Log Rank

3. Secondary Outcome: Percentage of Participants With Survival Idiopathic Pulmonary Fibrosis (IPF) -Related Mortality Events
Description: IPF-related mortality events were defined as deaths due to IPF related cause. Kaplan-Meier estimates of the percentage of participants with the event of interest along with 80% two-sided confidence intervals using Greenwood's formula are provided.
Time Frame: Up to 48 weeks post first dose of study treatment
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | VAY736 | Placebo
Number analyzed (Participants) | 12 | 16
Percentage of participants | 0 [NA to NA] — NA: Not estimable because no events occurred within this group | 0 [NA to NA] — NA: Not estimable because no events occurred within this group

4. Secondary Outcome: Percentage of Participants With Progression-free Survival (PFS) Events
Description: PFS events were divided into: 1) PFS1 events including progression (relative reduction in FVC ≥ 10%) or death due to all causes, and 2) PFS2 events including progression (relative reduction in FVC ≥ 10%) or death due to IPF-related causes. Kaplan-Meier estimates of the percentage of participants with the event of interest (PFS1 events or PFS2 events) along with 80% two-sided confidence intervals using Greenwood's formula are provided.
Time Frame: Up to 48 weeks post first dose of study treatment
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | VAY736 | Placebo
Number analyzed (Participants) | 12 | 16
Percentage of participants
  PFS1 | 61.0 [38.22 to 84.20] | 31.9 [18.04 to 52.51]
  PFS2 | 57.1 [33.44 to 82.86] | 31.9 [18.04 to 52.51]
Statistical Analysis 1: Comparison: VAY736 vs Placebo; PFS1; Test type: Other; p = 0.921, Log Rank; Hazard Ratio (HR) = 2.6, 80% CI 2-sided [1.1 to 6.3]
Statistical Analysis 2: Comparison: VAY736 vs Placebo; PFS2; Test type: Other; p = 0.863, Log Rank; Hazard Ratio (HR) = 2.2, 80% CI 2-sided [0.9 to 5.6]

5. Secondary Outcome: Percentage of Participants With Disease Progression Events
Description: The following disease progression events were considered: a) relative reduction in FVC ≥ 10%; b) relative reduction in Diffusing Capacity of the Lungs (DLCO) ≥ 15%; c) absolute reduction in Six Minute Walk Distance (6MWD) ≥ 50 m. Kaplan-Meier estimates of the percentage of participants with the event of interest along with 80% two-sided confidence intervals using Greenwood's formula are provided.
Time Frame: Up to 48 weeks post first dose of study treatment
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | VAY736 | Placebo
Number analyzed (Participants) | 12 | 16
Percentage of participants
  FVC | 57.1 [33.44 to 82.86] | 31.9 [18.04 to 52.51]
  DLCO | 73.8 [46.56 to 94.24] | 56.1 [38.65 to 75.10]
  6MWD | 38.3 [19.96 to 64.88] | 75.0 [58.52 to 88.74]
Statistical Analysis 1: Comparison: VAY736 vs Placebo; FVC; Test type: Other; p = 0.863, Log Rank; Hazard Ratio (HR) = 2.2, 80% CI 2-sided [0.9 to 5.6]
Statistical Analysis 2: Comparison: VAY736 vs Placebo; DLCO; Test type: Other; p = 0.457, Log Rank; Hazard Ratio (HR) = 0.9, 80% CI 2-sided [0.4 to 2.0]
Statistical Analysis 3: Comparison: VAY736 vs Placebo; 6MWD; Test type: Other; p = 0.019, Log Rank; Hazard Ratio (HR) = 0.3, 80% CI 2-sided [0.1 to 0.6]

6. Secondary Outcome: Percentage of Participants With Composite Events
Description: Composite events were defined as: 1) death (all-cause mortality), or relative reduction in FVC ≥ 10%, or relative reduction in DLCO ≥ 15%, or relative reduction in 6MWD ≥ 50 m (composite endpoint 1); and 2) Death (IPF-related mortality), or relative reduction in FVC ≥ 10%, or relative reduction in DLCO ≥ 15%, or relative reduction in 6MWD ≥ 50 m (composite endpoint 2). Kaplan-Meier estimates of the percentage of participants with the event of interest along with 80% two-sided confidence intervals using Greenwood's formula are provided.
Time Frame: Up to 48 weeks post first dose of study treatment
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | VAY736 | Placebo
Number analyzed (Participants) | 12 | 16
Percentage of participants
  Composite Endpoint 1 | 81.0 [63.86 to 93.29] | 66.3 [50.84 to 81.18]
  Composite Endpoint 2 | 79.2 [61.07 to 92.70] | 66.3 [50.84 to 81.18]
Statistical Analysis 1: Comparison: VAY736 vs Placebo; Composite Endpoint 1; Test type: Other; p = 0.611, Log Rank; Hazard Ratio (HR) = 1.1, 80% CI 2-sided [0.6 to 2.0]
Statistical Analysis 2: Comparison: VAY736 vs Placebo; Composite Endpoint 2; Test type: Other; p = 0.549, Log Rank; Hazard Ratio (HR) = 1.1, 80% CI 2-sided [0.6 to 1.9]

7. Secondary Outcome: Change From Baseline to End of Treatment Epoch (48 Weeks of Treatment) in Diffusing Capacity of the Lungs
Description: DLCO is a measurement to assess the lungs' ability to transfer gas from inspired air to the bloodstream. DLCO was determined according to ATS guidelines. Change from baseline to end of treatment epoch (48 weeks of treatment) in diffusing capacity of the lung for carbon monoxide (DLCO) was analyzed using a Mixed Effects Model for Repeated Measures (MMRM) and considering all assessments collected during the treatment epoch. The model included treatment and visit as fixed effects, standard of care treatment (Nintedanib, Pirfenidone, or no treatment) as factor and baseline value as a covariate, treatment-by-visit and baseline-by-visit as interaction terms. A positive change from baseline indicates improvement.
  Baseline was defined as the last available assessment pre-dose before or on randomization date.
Time Frame: From baseline up to 48 weeks post first dose of study treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mililiter/minute/millimeter Mercury
Arm/Group | VAY736 | Placebo
Number analyzed (Participants) | 3 | 7
mililiter/minute/millimeter Mercury | -1.954 (1.0816) | -1.033 (0.7244)
Statistical Analysis 1: Comparison: VAY736 vs Placebo; Test type: Superiority; p = 0.7576, MMRM — 1-sided p-values were obtained using MMRM Model; Least Squares of the Mean = -0.920, 80% CI 2-sided [-2.615 to 0.774], Standard Error of Mean 1.3109

8. Secondary Outcome: Change From Baseline to the End of Treatment Epoch (48 Weeks of Treatment) in 6-minute Walk Distance (6MWD)
Description: A standardized 6-minute walk test (6MWT) was performed in accordance with the guidelines of the American Thoracic Society 2002. The distance walked in six minutes (6MWD) was recorded. Change from baseline to end of treatment epoch (48 weeks of treatment) in 6MWD was analyzed using a Mixed Effects Model for Repeated Measures (MMRM) and considering all assessments collected during the treatment epoch. The model included treatment and visit as fixed effects, standard of care treatment (Nintedanib, Pirfenidone, or no treatment) as factor and baseline value as a covariate, treatment-by-visit and baseline-by-visit as interaction terms. A positive change from baseline indicates improvement. Baseline was defined as the last available assessment pre-dose before or on randomization date.
Time Frame: From baseline up to 48 weeks post first dose of study treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Meter (m)
Arm/Group | VAY736 | Placebo
Number analyzed (Participants) | 2 | 7
Meter (m) | 19.743 (53.5268) | -12.479 (28.9400)
Statistical Analysis 1: Comparison: VAY736 vs Placebo; Test type: Superiority; p = 0.3018, MMRM — 1-sided p-values were obtained using MMRM Model; Least Squares of the Mean = 32.222, 80% CI 2-sided [-47.572 to 112.015], Standard Error of Mean 61.8632

9. Secondary Outcome: Change From Baseline to the End of Treatment Epoch (48 Weeks of Treatment) in Distance Saturation Product
Description: Distance saturation product is the product of distance walked and lowest oxygen saturation during the 6-min walk test. Change from baseline to end of treatment epoch (48 weeks of treatment) in distance saturation product was analyzed using a Mixed Effects Model for Repeated Measures (MMRM) and considering all assessments collected during the treatment epoch. The model included treatment and visit as fixed effects, standard of care treatment (Nintedanib, Pirfenidone, or no treatment) as factor and baseline value as a covariate, treatment-by-visit and baseline-by-visit as interaction terms. A positive change from baseline indicates improvement. Baseline was defined as the last available assessment pre-dose before or on randomization date.
Time Frame: From baseline up to 48 weeks post first dose of study treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Meter% (m%)
Arm/Group | VAY736 | Placebo
Number analyzed (Participants) | 2 | 7
Meter% (m%) | 9.746 (52.2985) | -19.420 (28.3755)
Statistical Analysis 1: Comparison: VAY736 vs Placebo; Test type: Superiority; p = 0.3140, MMRM — 1-sided p-values were obtained using MMRM Model; Least Squares of the Mean = 29.166, 80% CI 2-sided [-48.220 to 106.553], Standard Error of Mean 60.0143

10. Secondary Outcome: Change From Baseline to the End of Treatment Epoch (48 Weeks of Treatment) in Resting Oxygen Saturation Level (on Room Air)
Description: Change from baseline to end of treatment epoch (48 weeks of treatment) in resting oxygen saturation (on room air) was analyzed using a Mixed Effects Model for Repeated Measures (MMRM) and considering all assessments collected during the treatment epoch. The model included treatment and visit as fixed effects, standard of care treatment (Nintedanib, Pirfenidone, or no treatment) as factor and baseline value as a covariate, treatment-by-visit and baseline-by-visit as interaction terms. A positive change from baseline indicates improvement. Baseline was defined as the last available assessment pre-dose before or on randomization date.
Time Frame: From baseline up to 48 weeks post first dose of study treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Arm/Group | VAY736 | Placebo
Number analyzed (Participants) | 5 | 7
Percentage (%) | -0.117 (1.0179) | -1.887 (0.9415)
Statistical Analysis 1: Comparison: VAY736 vs Placebo; Test type: Superiority; p = 0.1269, MMRM — 1-sided p-values were obtained using MMRM Model; Least Squares of the mean = 1.770, 80% CI 2-sided [-0.219 to 3.759], Standard Error of Mean 1.5422

11. Secondary Outcome: Number of Participants With Positive Serum Anti-VAY736 Antibodies
Description: Number of participants with positive serum anti-VAY736 antibodies. A bridging ELISA method that is designed to detect the presence of anti-VAY736 antibodies in human serum was used.
Time Frame: Day 1, 29, 85, 169, 253 and 337
Population: Immunogenicity (IG) analysis set including all participants with at least one available valid (i.e. not flagged for exclusion) IG concentration measurement, who received any study drug and with no protocol deviations that impact on IG data.
Measure: Number; unit: Participants
Arm/Group | VAY736 | Placebo
Number analyzed (Participants) | 10 | 15
Participants
  Day 1 | 1 | 3
  Day 29 | 1 | 2
  Day 85 | 1 | 1
  Day 169 | 0 | 2
  Day 253 | 2 | 1
  Day 337 | 0 | 0

12. Secondary Outcome: Ctrough of VAY736 From the Serum Concentration-time Data
Description: The lowest serum concentration of VAY736 observed during a dosing interval at steady state (Ctrough) was determined
Time Frame: At pre-dose on Day 1, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309 and 337
Population: Overall number of participants analyzed represents the Pharmacokinetic (PK) analysis set including all participants with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement who received at least one dose of VAY736 and with no protocol deviations that impact on PK data. The number of participants analyzed in each row represents the number of participants with a valid value in the corresponding time point.
Measure: Mean (Standard Deviation); unit: nanogram (ng) / mililiter (mL)
Arm/Group | VAY736
Number analyzed (Participants) | 11
nanogram (ng) / mililiter (mL)
  Day 1 | 0.00 (0.000)
  Day 29: number analyzed (Participants) | 8
  Day 29 | 676.79 (499.931)
  Day 57: number analyzed (Participants) | 9
  Day 57 | 779.89 (645.363)
  Day 85: number analyzed (Participants) | 8
  Day 85 | 786.63 (501.225)
  Day 113: number analyzed (Participants) | 8
  Day 113 | 771.88 (623.268)
  Day 141: number analyzed (Participants) | 6
  Day 141 | 1316.05 (877.240)
  Day 169: number analyzed (Participants) | 7
  Day 169 | 1019.00 (587.097)
  Day 197: number analyzed (Participants) | 4
  Day 197 | 985.50 (495.652)
  Day 225: number analyzed (Participants) | 4
  Day 225 | 1271.10 (863.055)
  Day 253: number analyzed (Participants) | 7
  Day 253 | 998.57 (947.343)
  Day 281: number analyzed (Participants) | 2
  Day 281 | 705.00 (997.021)
  Day 309: number analyzed (Participants) | 5
  Day 309 | 827.40 (678.836)
  Day 337: number analyzed (Participants) | 6
  Day 337 | 688.50 (1172.124)

ADVERSE EVENTS:
Time Frame: From baseline up to end of study, assessed up to approximately 2.4 years
Description: Safety analyses were performed in the safety set including all participants who received at least one dose of any study drug
Groups:
- Total: Total
Arm/Group | VAY736 | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/16 | 1/29
Serious Adverse Events (participants affected / at risk) | 5/13 | 9/16 | 14/29
Other Adverse Events (participants affected / at risk) | 13/13 | 15/16 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAY736 (N=13) | Placebo (N=16) | Total (N=29)
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Vasculitis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VAY736 (N=13) | Placebo (N=16) | Total (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Corneal degeneration (Eye disorders) | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3
Asthenia (General disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 3
Injection site bruising (General disorders) | 1 | 1 | 2
Injection site dermatitis (General disorders) | 1 | 0 | 1
Injection site erythema (General disorders) | 2 | 1 | 3
Injection site inflammation (General disorders) | 1 | 0 | 1
Injection site pain (General disorders) | 0 | 1 | 1
Injection site pruritus (General disorders) | 3 | 2 | 5
Injection site rash (General disorders) | 1 | 0 | 1
Injection site warmth (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 2 | 4
Conjunctivitis (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Respiratory tract infection (Infections and infestations) | 2 | 1 | 3
Rhinitis (Infections and infestations) | 0 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 4
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 2
Sunburn (Injury, poisoning and procedural complications) | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 2 | 0 | 2
Antinuclear antibody increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase decreased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 1
Blood parathyroid hormone decreased (Investigations) | 1 | 0 | 1
Blood potassium increased (Investigations) | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 1
Blood urea increased (Investigations) | 1 | 0 | 1
Blood urine present (Investigations) | 1 | 0 | 1
Escherichia test positive (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 2
Glucose urine present (Investigations) | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 1
Mean cell volume increased (Investigations) | 1 | 0 | 1
Monocyte count increased (Investigations) | 2 | 0 | 2
Neutrophil count increased (Investigations) | 1 | 0 | 1
Protein urine present (Investigations) | 0 | 1 | 1
Urine albumin/creatinine ratio increased (Investigations) | 0 | 1 | 1
Urine analysis abnormal (Investigations) | 1 | 0 | 1
Urine protein/creatinine ratio increased (Investigations) | 1 | 1 | 2
Weight decreased (Investigations) | 1 | 4 | 5
White blood cell count increased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 2 | 4
Memory impairment (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 1 | 3
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Keloid scar (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hot flush (Vascular disorders) | 2 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT03287414/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT03287414/SAP_001.pdf